CLINICAL TRIAL: NCT01336855
Title: Collection and Preservation of Blood and Serum Specimens From HIV Positive or HIV Negative Patients for Multiple Collaborative Studies
Brief Title: Collection of Blood for Multiple Collaborative Studies
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H8211-04743-22
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: HIV
Keywords: HIV; Observational; Pathogenesis; Immunology; Virology; Control; Healthy control; Men who have sex with men
MeSH Terms: conditions — Homosexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, PBMCs, buffy coat, serum, saliva, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HIV Positive: HIV-1 positive subjects
- HIV negative subjects: HIV-1 seronegative control group

SUMMARY:
This study seeks to confidentially collect blood from HIV-positive individuals and HIV-negative controls to provide basic scientists with specimens for collaborative studies.

DETAILED DESCRIPTION:
HIV positive patients are currently the focus of multiple collaborative research studies, both at UCSF and other institutions. The aims of these research projects include improving the understanding of etiology, immunology, epidemiology and treatment of HIV. There are numerous requests from basic scientists at UCSF for collaborative studies on specimens, especially for blood, saliva and urine samples. Specimens may be used to test such things as virus characteristics, genotyping and/or phenotyping resistance, plasma drug concentrations, immune function or evidence of complications of HIV disease. The samples may also be tested for genetic factors that may be related to the course of HIV disease

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 antibody negative with similar characteristics to HIV-1 positive cohort
* HIV-positive subjects naive to antiretroviral therapy
* HIV-positive subjects stable on or off antiretroviral therapy for a minimum of 6 months
* Good venous access
* Able to provide informed consent

Exclusion Criteria:

* Hemoglobin < 9g/dl
* Hematocrit < 27%
* Active treatment for cancer
* Hospitalization or IV antibiotic use within the last 4 months
* Immunosuppressive therapy within the last 4 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected based on positive or negative HIV antibody, depending on the study for which blood is being collected. Patients will be chosen from the Positive Health Practice populations at SFGH and UCSF, the General Medicine Clinic at the San Francisco Veterans Affairs Medical Center. HIV uninfected healthy volunteers with comparable risk factors to the HIV positive subjects will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1988-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Plasma HIV RNA level | Ongoing
  Viral load

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, M.D., Principal Investigator — University of Californa, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No